CLINICAL TRIAL: NCT01105741
Title: Metabolomic Analysis, a Potential Tool to Direct Treatment With Adalimumab in Crohn's Disease (CD)
Acronym: MB
Status: Completed | Type: Observational
Sponsor: Martin Storr (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Martin Storr, MD, University of Calgary
Organization: University of Calgary (Other)
Other Study IDs: E-22684
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Adalimumab; Metabolome
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Active Crohn's disease - single arm: Active Crohn's disease, a decision is made to start treatment with adalimumab.

SUMMARY:
Background and Rationale: Inflammatory bowel disease (IBD) is a major burden to individuals and society. Ulcerative colitis and Crohn's disease (CD) are the 2 major inflammatory bowel diseases (IBD). They share some pathologic and clinical features but overall their pathogenesis is not resolved and diagnosis is sometimes difficult. The incidence rates range from 3.1 to 14.6 cases per 100,000 person year for Crohn's disease to 2.2 to 14.3 cases per 100,000 person years for ulcerative colitis and prevalence ranges up to 201/100,000 for Crohn's disease and up to 246/100,000 persons for ulcerative colitis.

Powerful biological therapies were recently introduced for the treatment of CD. They offer superior treatment for the treatment of steroid refractory patients. Interestingly newer studies suggest that these therapies might also be beneficial if not superior if used at earlier stages of the disease. But presently limitations of these treatments need to be considered and biomarkers that could better direct these treatments are urgently needed.

One present limitation is that these new therapies, though being beneficial in a large number of CD patients, will not be beneficial to all CD patients. Presently treatment responders and non-responders can not be identified prior to the treatment with the biological adalimumab representing an important unmet clinical need. Since adalimumab treatment can be accompanied by serious, potentially lethal, side effects, it would be a major advantage if future biomarkers could predict whether an individual will or will not respond to one or the other treatment.

Furthermore with treatments available being associated with high costs to patients and society, as the treatment with adalimumab is, biomarkers that would help to identify potential treatment-responders or non-responders would support their targeted use and would be appreciated by all stakeholders.

Nuclear magnetic resonance (NMR) spectroscopy is a method that generates comprehensive metabolic profiles from human biofluids, and these metabolomic profiles may be useful to identify biomarkers with discriminative and predictive power in CD. Thereby amongst other factors serum metabolites are affected by inflammation and urine metabolites are affected by gut flora and thus one or a combination of both may be a valuable tool in CD.

Aim: The investigators aim is to identify metabolomic predictors of clinical response to adalimumab treatment in CD patients in order to direct future treatment to a group of patients that is expected to benefit most.

Methods: Metabolomic profiling together with the collection of clinical data will be performed in patients with IBD prior to treatment with biological therapy and for up to 6 month thereafter.

In the study the investigators follow 50 patients with Crohn's Disease, naive to treatment with biologics. Metabolomic profiling will be performed 1 week prior to the treatment with adalimumab and then every 4 weeks for 6 month. In order to be reliable and reproducible, sampling will be performed in the morning after an overnight fasting period. On the days of serum/urine collection the following data will be collected: CBC, ESR, CRP, Calprotectin, ASCA/pANCA, IL-10, TNFα, IFNγ, Crohn's disease Activity Index, present medication and OTC, Dietary and lifestyle history including 24 hour dietary recall, alcohol intake, smoking and exercise.

Multivariate analysis will be performed to identify patterns in the metabolomic profile that predict response or non-response to adalimumab treatment.

To summarize, IBD is a major burden to patients and society. Adalimumab treatment is helpful in steroid refractory patients. Novel biomarkers that help physicians to decide which patient might benefit from adalimumab treatment may be powerful tools to optimize directing these powerful but expensive and side effect bearing therapies towards the patient that might benefit most. Metabolomic profiling may be the tool that helps us to identify these patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject has active Crohn's disease (as determined by treating gastroenterologist)
* Age ≥ 18 years old
* Commencing treatment with adalimumab according to product label (at the discretion of their responsible gastroenterologist)
* Willing to attend scheduled protocol visits, complete required study procedures and able to fast overnight
* No previous treatment with anti-TNF therapies or other biological therapies (i.e., cytokines), including investigational agents

Exclusion Criteria:

* Subject has inactive Crohn's disease (as determined by treating gastroenterologist)
* Indeterminate colitis or Ulcerative colitis
* Age < 18 years old
* Previous or present treatment with a biological (anti-TNF therapies, cytokines), including investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's disease, active disease
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Treatment successfully defined by decrease of Disease Activity Index (DAI) of 3 or more at week 24 | 24 weeks

SECONDARY OUTCOMES:
changes in metabolomic profile | 24 weeks
  The metabolic profil consists of 75 metabolites. These metabolites will be measured and changes will be captured.
Change in CRP | 24 weeks
  CRP will be measured in blood serum
change in medication use | 24 weeks
  Medication use will be recorded on every visit, changes in use will be captured.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Storr, MD, Principal Investigator — University Calgary; Martin Storr, MD, Study Director — University Calgary
Locations (1):
- Division of Gastroenterology, Calgary, Alberta, Canada